CLINICAL TRIAL: NCT03983304
Title: Electromagnetic Muscle Stimulation for Abdominal and Gluteal Muscle Toning
Brief Title: EMS for Abdominal and Gluteal Muscle Toning
Acronym: CTP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZA19-002
Record Dates: First submitted 2019-06-10; First posted 2019-06-12 (Actual); Results first posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Non-Therapeutic Body Modification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Electromagnetic Muscle Stimulation Treatment Group - Abdomen (Experimental): The treatments are designed to evaluate muscle toning, firming and strengthening in the abdomen.
  Interventions: Device: The ZELTIQ EMS System
- Electromagnetic Muscle Stimulation Group - Abdomen and Buttocks (Experimental): The treatments are designed to evaluate muscle toning, firming and strengthening in the abdomen and buttocks.
  Interventions: Device: The ZELTIQ EMS System

INTERVENTIONS:
Device: The ZELTIQ EMS System — The Zeltiq EMS device will be used to perform treatments for abdominal and gluteal toning.

SUMMARY:
Evaluate the use of Electromagnetic Muscle Stimulation for body contouring.

DETAILED DESCRIPTION:
The safety and effectiveness of an Electromagnetic Muscle Stimulation device when used for abdominal and gluteal toning will be evaluated in this study.

ELIGIBILITY:
Inclusion Criteria

* Male or female ≥ 22 years and ≤65 years of age.
* Subject has not had weight change exceeding 5% of body weight in the preceding month.
* Subject agrees to maintain body weight within 5% during the study by not making any changes in diet or exercise routine.
* Subject has a BMI ≤ 30 as determined at screening.
* Subject agrees to have photographs taken of the treatment area(s) during the scheduled time periods.
* Subject agrees to refrain from any new abdominal and/or gluteal muscle training exercises of the treatment area during the course of the study.
* Subject agrees to avoid sun tanning during the course of the study.
* Subject has read and signed the study written informed consent form.

Exclusion Criteria

* Subject has had a recent surgical procedure(s) in the area of intended treatment and muscle contractions may disrupt the healing process.
* Subject has had an invasive fat reduction procedure (e.g., liposuction, mesotherapy) in the area of intended treatment.
* Subject needs to administer or has a known history of subcutaneous injections into the area of intended treatment (e.g., heparin, insulin) within the past month.
* Subject has not had an intrauterine contraceptive device inserted or removed within the past month.
* Subject has a bleeding disorder
* Subject is taking or has taken diet pills or supplements within the past month.
* Subject has a metal implant or active implanted device such as a cardiac pacemaker, cochlear implant, intrathecal pump, hearing aids, defibrillator, or drug delivery system.
* Subject agrees not to change muscle exercise routine in the treatment area (abdominal and/or gluteal) while participating in the study
* Subject has pulmonary insufficiency.
* Subject has a cardiac disorder.
* Subject has a malignant tumor.
* Subject has been diagnosed with a seizure disorder such as epilepsy.
* Subject currently has a fever.
* Subject is diagnosed with Grave's disease.
* Subject is pregnant or intending to become pregnant during the study period (in the next 9 months).
* Subject is lactating or has been lactating in the past 6 months.
* Subject is unable or unwilling to comply with the study requirements.
* Subject is currently enrolled in a clinical study of any other investigational drug or device.
* Any other condition or laboratory value that would, in the professional opinion of the Investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerrie Jiang, NP, Study Director — Zeltiq Aesthetics
Locations (8):
- United States (8):
  - Marina Plastic Surgery, Marina del Rey, California
  - Innovation Research Center, Pleasanton, California
  - Cosmetic Laser Dermatology, San Diego, California
  - Bowes Dermatology by Riverchase, Miami, Florida
  - The Wall Center for Plastic Surgery, Shreveport, Louisiana
  - Capital Laser & Skin Care, Chevy Chase, Maryland
  - SkinCare Physicians of Chestnut Hill, Chestnut Hill, Massachusetts
  - EpiCentre Park Lane, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fabi S, Dover JS, Tanzi E, Bowes LE, Tsai Fu F, Odusan A. A 12-Week, Prospective, Non-Comparative, Non-Randomized Study of Magnetic Muscle Stimulation for Improvement of Body Satisfaction With the Abdomen and Buttocks. Lasers Surg Med. 2021 Jan;53(1):79-88. doi: 10.1002/lsm.23348. Epub 2020 Nov 8. PMID 33161584

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants received EMS therapy on abdomen and/or buttocks in 4 sessions over a 2-week period, with follow-up visits 4 and 12 wks post final treatment. Per-protocol Population included all treated participants followed for 4 wks post treatment, with weight change of no more than 5% of total body weight at the time of the 4-Wk post-treatment images compared to baseline (pre-treatment) images, and who completed 4 treatments. Per protocol, data presented here as planned/collected (all enrolled).
Groups:
- EMS Device Treatment Group: All enrolled participants treated with the EMS device.
Period: Overall Study
Arm/Group | EMS Device Treatment Group
Started | 110
Completed | 103
Not Completed | 7
Not completed — Withdrawal by Subject | 5
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Data presented here as planned and collected (all enrolled).
Arm/Group | EMS Device Treatment Group
Number analyzed (Participants) | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 110
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83
  Male | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Am Indian or Alaska Native | 0
  Asian | 9
  Black or African American | 4
  Native Hawaiian or Pac Islander | 0
  White | 88
  Other | 8
  Unknown - Missing Data Point | 1
Region of Enrollment [Number; unit: participants]
  United States | 110
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.3 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Satisfaction Questionnaire From Baseline to 4-Week Post-Treatment Follow-up Visit
Description: Measurement of participant's perception about body shape, assessed using the Body Satisfaction Questionnaire (BSQ)at the 4-Week post-treatment follow-up visit. The scale measures body image using a set of dichotomous items used to describe aspects of shape and appearance. The questionnaire has total score range from 10 to 50. An increase in score (when compared to baseline) reflects the participant's perceived improvement in appearance in the treated region(abdomen or buttocks). Questionnaire results were tabulated as the numerical change between mean baseline scores and scores recorded at the 4-week post-treatment follow-up visit. A positive change reflects an increase in the body satisfaction questionnaire total score.
Time Frame: Baseline, 4-week post-treatment follow-up visit
Population: Per-protocol population. Participants with completed questionnaires specific to each body area treated.
Measure: Mean (Standard Deviation); unit: Participants completed Questionnaire
Groups:
- EMS Device Treatment - Abdomen: All eligible participants for whom informed consent is obtained will be treated on the abdomen with the study device, an electromagnetic muscle stimulation device.
- EMS Treatment - Buttocks: All eligible participants for whom informed consent is obtained will be treated on the buttocks with the study device, an electromagnetic muscle stimulation device.
Arm/Group | EMS Device Treatment - Abdomen | EMS Treatment - Buttocks
Number analyzed (Participants) | 92 | 32
Participants completed Questionnaire | 5.1 (5.4) | 5.5 (5.3)

2. Primary Outcome: Number of Incidents of Device-Related Adverse Events
Description: The incidence of device-related adverse events (AE) including device-related serious AEs will be tabulated.
Time Frame: AE information will be collected from the time of enrollment to the final follow-up visit at 12 weeks following the final treatment.
Population: All participants enrolled in the study and treated with the EMS device were evaluated for adverse events throughout the study. Investigators determined if an AE was not related, possibly related, probably related or definitely related to the study device. Data is presented here as planned and collected per protocol, by the total As-Treated Population (defined as all treated participants regardless of weight change).
Measure: Number; unit: Device-Related Adverse Events
Groups:
- EMS Device Treatment Group: All eligible subjects for whom informed consent is obtained will be treated with the study device, an electromagnetic muscle stimulation device.
Arm/Group | EMS Device Treatment Group
Number analyzed (Participants) | 110
Device-Related Adverse Events | 6

3. Secondary Outcome: Percentage of Participants Reporting Improvement on the Subject Global Aesthetic Improvement Scale (SGAIS)
Description: Subject-graded improvement in the treated area using the Subject Global Aesthetic Scale (SGAIS) at the 4-Week follow-up visit. In this study, subjects completed the SGAIS questionnaire for each treated area (e.g. a abdomen-specific questionnaire and a buttocks-specific questionnaire) at the 4-week post-final follow-up visit. Subjects were asked to rate improvement in treated areas using the following 7 point scale:
  3 = Very much improved, 2 = Much improved, 1 = Improved, 0 = No change, -1 = Worse, -2 = Much worse and -3 = Very much worse. Subjects who reported 'Very Much Improved,' 'Much Improved,' and 'Improved will be categorized as 'Improved'. Results were calculated as the percentage of subjects reporting "Improved".
Time Frame: 4-week post-treatment follow-up visit
Population: Per-protocol population. Participants with completed questionnaires at the 4-week post treatment follow-up visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- EMS Treatment Device - Abdomen Questionnaire: Participants treated on the abdomen with the EMS device completed Subject Global Improvement Scale questionnaires at the 4-week follow-up visit.
- EMS Treatment Device - Buttocks: Participants treated on the buttocks with the EMS device completed Subject Global Improvement Scale questionnaires at the 4-week follow-up visit.
Arm/Group | EMS Treatment Device - Abdomen Questionnaire | EMS Treatment Device - Buttocks
Number analyzed (Participants) | 94 | 33
percentage of participants | 68.1 [57.7 to 77.3] | 81.8 [64.5 to 93.0]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the time of enrollment through the 12-week post-treatment follow-up visit, approximately 4 months.
Description: Safety data is presented here as planned and collected per protocol, by the total As-Treated Population (defined as all treated participants regardless of weight change).
Groups:
- EMS Device Treatment Group: All eligible subjects for whom informed consent is obtained were treated with the study device, an electromagnetic muscle stimulation device. Adverse event information was collected from the time of enrollment through the 12-week post-treatment follow-up visit.
  Per protocol 110 subjects were enrolled to have EMS treatments on the abdomen and/or buttocks in this single arm study. At no point in the conduct of the study were subjects assigned to a treatment group; the investigator determined the area(s) to be treated.
Arm/Group | EMS Device Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/110
Serious Adverse Events (participants affected / at risk) | 1/110
Other Adverse Events (participants affected / at risk) | 11/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EMS Device Treatment Group (N=110)
Lymphoma (Blood and lymphatic system disorders) | 1 (1) — Subject reported pain in the abdomen and other symptoms. Investigator referred subject to primary care physician. Subject diagnosed with lymphoma 18 days after treatment. Investigator determined the event as "not related to the study device.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EMS Device Treatment Group (N=110)
Elective surgery (Surgical and medical procedures) | 1 (1) — Subject reported elective salivary gland surgery.
Uterine Fibroid (Reproductive system and breast disorders) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Coughing (General disorders) | 1 (1)
Cold (virus) (General disorders) | 1 (1)
Sprained ankle (Musculoskeletal and connective tissue disorders) | 1 (1)
Menstrual Cycle Irregularity (General disorders) | 4 (4)
Soreness and discomfort in left chest (General disorders) | 1 (1)
Cramping in lower abdomen (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-10): https://cdn.clinicaltrials.gov/large-docs/04/NCT03983304/Prot_SAP_000.pdf